CLINICAL TRIAL: NCT06696976
Title: Effects of Telerehabilitation Versus Clinical Rehabilitation on Neuropathic Pain, Physical Function and Quality of Life in Chemotherapy Induced Peripheral Neuropathy
Brief Title: Effects of Telerehabilitation Versus Clinical Rehabilitation on Chemotherapy Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0229
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy
Keywords: Chemotherapy induced peripheral neuropathy; Telerehabilitation; Quality of life
MeSH Terms: interventions — Telerehabilitation; Treatment Outcome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (telerehabilitation of neuropathic pain, physical function and quality of life) (Experimental): Group A will receive Telerehabilitation of 60 minutes with short resting intervals .Treatment will be given 3 times per week for 12 weeks.
  1. warm up of 5 minutes
  2. Nerve gliding exercises of 10 minutes
  3. Balance exercises of 20 minutes
  4. Resistance training of 20 minutes
  5. cold down of 5 minutes
  Interventions: Other: Telerehabilitation
- Group B (clinical rehabilitation of neuropathic pain, physical function and quality of life) (Experimental): Group B will receive Clinical rehabilitation of 60 minutes with short resting intervals .Treatment will be given 3 times per week for 12 weeks.
  1. warm up of 5 minutes
  2. Nerve gliding exercises of 10 minutes
  3. Balance exercises of 20 minutes
  4. Resistance training of 20 minutes
  5. cold down of 5 minutes
  Interventions: Other: Clinical rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — A qualified physiotherapist himself used the digital platform Zoom (Zoom Video Communications or WhatsApp video communication) to deliver synchronic online sessions (60 min each), sending each participant a link by email, half an hour before the weekly meetings. The patients were also invited to present themselves in comfortable gymnastic clothing and with tools useful for the motor program: a chair, a stick, a bottle full of water (or small weights if the patient had them), and a mat.
  Nerve gliding exercises: These 5 Nerve gliding exercises will perform 3 times a week requiring 10 minutes to complete.
  Balance exercises: Balance exercise include 10 exercises and take 20 minutes of completion, 2minute for each exercise.
  Resistance training using Thera Band will performed with the presence of the researcher as an instructor.The main upper-extremity movements consisted of chest press, shoulder press etc and in lower extremity such as leg press ,back thgh press etc. in patient.
  Arms: Group A (telerehabilitation of neuropathic pain, physical function and quality of life)
Other: Clinical rehabilitation — A qualified physiotherapist himself used the digital platform Zoom (Zoom Video Communications or WhatsApp video communication) to deliver synchronic online sessions (60 min each), sending each participant a link by email, half an hour before the weekly meetings. The patients were also invited to present themselves in comfortable gymnastic clothing and with tools useful for the motor program: a chair, a stick, a bottle full of water (or small weights if the patient had them), and a mat.
  Nerve gliding exercises: These 5 Nerve gliding exercises will perform 3 times a week requiring 10 minutes to complete.
  Balance exercises: Balance exercise include 10 exercises and take 20 minutes of completion, 2minute for each exercise.
  Resistance training using Thera Band will performed with the presence of the researcher as an instructor.The main upper-extremity movements consisted of chest press, shoulder press etc and in lower extremity such as leg press ,back thgh press etc. in patient.
  Arms: Group B (clinical rehabilitation of neuropathic pain, physical function and quality of life)

SUMMARY:
The aim of this study is to determine the comparative effects of telerehabilitation versus clinical rehabilitation on neuropathic pain, physical function and quality of life in Chemotherapy induced peripheral neuropathy patients.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is among the most prevalent and debilitating adverse effects of cancer treatment. CIPN increase risk of falls and impair physical function and quality of life (QOL). Physical therapy improves the CIPN symptoms, quality of life and physical function in cancer patients after chemotherapy. Telerehabilitation technologies such as telephone and video conferencing, have the capability of bringing services into the survivors' home and manage the symptoms without needing to have direct physical contact with the hospital or clinic services. The aim of this study is to determine the comparative effects of telerehabilitation versus clinical rehabilitation on neuropathic pain, physical function and quality of life.

This study will be a randomized clinical trial that will conducted at Gujranwala institute of Nuclear Medicine hospital in which sixty-six cancer patient who will sustain grade 3 and grade 4 of European Organization for Research and Treatment of Cancer Quality of life-Chemotherapy Induced Peripheral Neuropathy Questionnaire (EORTC-QLQ-CIPN20)will randomly allocated to Group A(n=33)who will receive Telerehabilitation and Group B (n=33) who will receive clinical rehabilitation using the computer generated method. The sample size calculated for this trial will be 66. Interventions will be given in both groups for 60 minutes for 12 weeks (3times per week).10 minutes for Nerve Gliding exercises ,20 minutes for Balance training and 20 minutes forResistance training (using Therapeutic band).European Organization for Research and Treatment of Cancer Quality of Life-Chemotherapy Induced Peripheral Neuropathy Questionnaire (EORTC QLQ-CIPN20) will be used to assess quality of life. Berg balance scale for balance and Manual Muscle testing for muscle strength. The data will be entered and analyzed using SPSS 26. Statistical significance will be set at p=0.05. Normality of data will be assessed through Kolmogorov-Smirnov test. Assessment will be carried out at baseline,6th week, 12th week after discontinuation of treatment and 18th week follow up. For between group analysis of parametric data Independent T test will be used, while Mann Whitney test will be applied for non-parametric data. For within group comparison repeated measure ANOVA will be used, for non-parametric data, Friedman ANOVA will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with breast cancer.
* Patients of age between 45 to 75years.
* Patient expected to survive for 6 month or more.
* Patient after specific chemotherapy such as taxanes(paclitaxel),vinca alkaloids(vinorelbine),bortezomib, lenalidomide and platinum-based.
* Patient with Stage 1 to 3.
* Patients have prior history of mechanical nerve entrapment without clinical symptoms (carpal tunnel syndrome) were included.
* Patient who sustained grade 3 and 4 of European Organization for Research and Treatment of Cancer Quality of Life-Chemotherapy-Induced Peripheral Neuropathy Questionnaire (EORTC QLQ-CIPN20).

Exclusion Criteria:

* Patients with history of peripheral neuropathy.
* Participants are excluded if they had comorbid conditions causing peripheral neuropathic symptoms (including previous chemotherapy or diabetes or alcohol abuse and non-alcoholic liver diseases.
* Patients not scheduled for one of the aforementioned taxane-based regimens.
* Patients with vitamin D or B12 deficiency.
* Non-ambulatory Patients.
* Patients reluctant to practice exercise program.
* Patient have impaired visual or vestibular system and presence of bone or any kind of central nervous system involvement , including cancer.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with breast cancer patient
Enrollment: 66 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE | 12th week
  Numeric Pain Rating Scale (NPRS) rated CIPN pain. The NPRS is an 11point scale (0-10) ranking pain from 0, indicating no pain at all, to 10, indicating worst pain imaginable on each assessment visit, of the finger tips. This was to identify pain specific to CIPN. A change score of 2 is reported to be a clinically relevant change. The numeric pain rating scale was used for pain measurement , the reliability of which is reported to be between 85% and 95%.
EORTC CIPN20 | 12th week
  The EORTC CIPN20 should provide valuable information on CIPN-related symptoms and functional limitations of patients exposed to potentially neurotoxic chemotherapeutic and/or neuroprotective agents. The resulting 20-item questionnaire was pre-tested in three languages and four countries and is currently being examined in a large, international clinical trial. The Chinese version of the EORTC QLQ-CIPN20 demonstrated acceptable reliability, validity and responsiveness and was found comparable in measuring CIPN among Chinese cancer patients.The questionnaire consists of sensory and motor neuropathy scales, autonomic scales for dizziness, blurred vision, and erectile dysfunction. The results obtained were converted into a 0-100 scale, with higher results indicating a higher degree of peripheral neuropathy.
The Berg balance scale (BBS): | 12th week
  Is considered the criterion standard in functional balance evaluation. In total, 14 different activities are scored between 0 (worst) and 4 (best), according to the patient's performance. The maximum score is 56. A total score close to 56 indicates that the balance of the patient is good, and lower scores denote poor balance established the validity and reliability of the Turkish version of the BBS.
Manual Muscle testing (MMT) | 12th week
  Is the most commonly used method for documenting impairments in muscle strength. Because of the variability possible during MMT, several studies examining MMT have used specialized instrumentation to provide support for the extremity tested and for standardization of joint position. Throughout its history manual muscle testing has been performed by practitioners' hands. Lamb states (1985) that MMT has content validity because the test construction is based on known physiologic, anatomic and kinesiologic principles. A number of research papers have dealt with this specific aspect of MMT in the diagnosis of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Phd, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Postma TJ, Aaronson NK, Heimans JJ, Muller MJ, Hildebrand JG, Delattre JY, Hoang-Xuan K, Lanteri-Minet M, Grant R, Huddart R, Moynihan C, Maher J, Lucey R; EORTC Quality of Life Group. The development of an EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy: the QLQ-CIPN20. Eur J Cancer. 2005 May;41(8):1135-9. doi: 10.1016/j.ejca.2005.02.012. Epub 2005 Apr 14. PMID 15911236
- [Background] Cheville AL, Moynihan T, Herrin J, Loprinzi C, Kroenke K. Effect of Collaborative Telerehabilitation on Functional Impairment and Pain Among Patients With Advanced-Stage Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):644-652. doi: 10.1001/jamaoncol.2019.0011. PMID 30946436
- [Background] Loubani K, Schreuer N, Kizony R. Telerehabilitation for Managing Daily Participation among Breast Cancer Survivors during COVID-19: A Feasibility Study. J Clin Med. 2022 Feb 16;11(4):1022. doi: 10.3390/jcm11041022. PMID 35207294
- [Background] van Egmond MA, Engelbert RHH, Klinkenbijl JHG, van Berge Henegouwen MI, van der Schaaf M. Physiotherapy With Telerehabilitation in Patients With Complicated Postoperative Recovery After Esophageal Cancer Surgery: Feasibility Study. J Med Internet Res. 2020 Jun 9;22(6):e16056. doi: 10.2196/16056. PMID 32515742
- [Background] Galiano-Castillo N, Arroyo-Morales M, Lozano-Lozano M, Fernandez-Lao C, Martin-Martin L, Del-Moral-Avila R, Cantarero-Villanueva I. Effect of an Internet-based telehealth system on functional capacity and cognition in breast cancer survivors: a secondary analysis of a randomized controlled trial. Support Care Cancer. 2017 Nov;25(11):3551-3559. doi: 10.1007/s00520-017-3782-9. Epub 2017 Jun 22. PMID 28639097
- [Background] Cottrell MA, O'Leary SP, Swete-Kelly P, Elwell B, Hess S, Litchfield MA, McLoughlin I, Tweedy R, Raymer M, Hill AJ, Russell TG. Agreement between telehealth and in-person assessment of patients with chronic musculoskeletal conditions presenting to an advanced-practice physiotherapy screening clinic. Musculoskelet Sci Pract. 2018 Dec;38:99-105. doi: 10.1016/j.msksp.2018.09.014. Epub 2018 Oct 4. PMID 30366292
- [Background] Dhawan S, Andrews R, Kumar L, Wadhwa S, Shukla G. A Randomized Controlled Trial to Assess the Effectiveness of Muscle Strengthening and Balancing Exercises on Chemotherapy-Induced Peripheral Neuropathic Pain and Quality of Life Among Cancer Patients. Cancer Nurs. 2020 Jul/Aug;43(4):269-280. doi: 10.1097/NCC.0000000000000693. PMID 30888982
- [Background] Zhang YH, Hu HY, Xiong YC, Peng C, Hu L, Kong YZ, Wang YL, Guo JB, Bi S, Li TS, Ao LJ, Wang CH, Bai YL, Fang L, Ma C, Liao LR, Liu H, Zhu Y, Zhang ZJ, Liu CL, Fang GE, Wang XQ. Exercise for Neuropathic Pain: A Systematic Review and Expert Consensus. Front Med (Lausanne). 2021 Nov 24;8:756940. doi: 10.3389/fmed.2021.756940. eCollection 2021. PMID 34901069
- [Background] Zimmer P, Trebing S, Timmers-Trebing U, Schenk A, Paust R, Bloch W, Rudolph R, Streckmann F, Baumann FT. Eight-week, multimodal exercise counteracts a progress of chemotherapy-induced peripheral neuropathy and improves balance and strength in metastasized colorectal cancer patients: a randomized controlled trial. Support Care Cancer. 2018 Feb;26(2):615-624. doi: 10.1007/s00520-017-3875-5. Epub 2017 Sep 30. PMID 28963591
- [Background] Stubblefield MD, McNeely ML, Alfano CM, Mayer DK. A prospective surveillance model for physical rehabilitation of women with breast cancer: chemotherapy-induced peripheral neuropathy. Cancer. 2012 Apr 15;118(8 Suppl):2250-60. doi: 10.1002/cncr.27463. PMID 22488699
- [Background] Mols F, Beijers T, Vreugdenhil G, van de Poll-Franse L. Chemotherapy-induced peripheral neuropathy and its association with quality of life: a systematic review. Support Care Cancer. 2014 Aug;22(8):2261-9. doi: 10.1007/s00520-014-2255-7. Epub 2014 May 1. PMID 24789421
- [Background] Bahar-Ozdemir Y, Akyuz G, Kalkandelen M, Yumuk PF. The Effect of Therapeutic Exercises on Balance, Quality of Life, and Pain in Patients Who Were Receiving Neurotoxic Chemotherapy. Am J Phys Med Rehabil. 2020 Apr;99(4):291-299. doi: 10.1097/PHM.0000000000001324. PMID 31592877